CLINICAL TRIAL: NCT07369960
Title: Randomized, Double-Blind Controlled Study for Transcranial Magnetic Stimulation Combined With Language Training in Children With Language Disorders in the Context of Global Developmental Delay
Brief Title: Transcranial Magnetic Stimulation Combined With Language Training for Language Disorders in Global Developmental Delay
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: Xiangxi Autonomous Prefecture People's Hospital (Unknown)
Responsible Party: Principal Investigator, shenwailiufangkun, Assistant Researcher, Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EC-LCKY2025078
Record Dates: First submitted 2026-01-06; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Transcranial Magnetic Stimulation; Language Disorders in Children; Developmental Delay Disorder
MeSH Terms: conditions — Developmental Disabilities | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcranial magnetic stimulation (Experimental): Receiving "true" high-frequency repetitive transcranial magnetic stimulation and personalized language training
  Interventions: Behavioral: Transcranial magnetic stimulation
- Control group (Sham Comparator): Receiving simulated pseudo-stimulation and personalized language training
  Interventions: Behavioral: Transcranial magnetic stimulation

INTERVENTIONS:
Behavioral: Transcranial magnetic stimulation — One group of children received non-invasive, painless magnetic stimulation therapy to activate the brain's language centers alongside personalized language training. Another group received identical-looking sham magnetic stimulation combined with personalized language training for scientific comparison. The entire study will last approximately 1 months, including 2 weeks of treatment and 2 weeks of follow-up

SUMMARY:
This study explores a safe and effective new approach to assisting children with Global Developmental Delay (GDD) and comorbid language disorders. Conducted at Xiangxi Autonomous Prefecture People's Hospital, the study will recruit approximately 50 children aged 2 to 5 years. Participants will be randomly assigned to one of two groups: one receiving personalized language training combined with non-invasive, painless repetitive Transcranial Magnetic Stimulation (rTMS) to activate language regions of the brain, and a control group receiving personalized training alongside sham stimulation for comparative analysis. The study spans one month, including a two-week intervention period followed by a two-week follow-up to evaluate the efficacy and sustainability of the combined therapy. This study has been rigorously reviewed and approved by the hospital's Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 2-5 years old, regardless of gender.
2. Meet the diagnostic definition of GDD in China's Diagnostic Guidelines for Global Developmental Delay (2024), confirmed by Gesell Developmental Schedules (GDS), and the Developmental Quotient (DQ) of the language domain is ≤75. At least one other of the four developmental domains, adaptive behavior, personal-social behavior, gross motor, and fine motor, had a DQ ≤ 75. Mild-moderate GDD was selected for the study.
3. The presence of significant language developmental delay, the language ability is significantly lower than children of the same age and the same intellectual level, confirmed by the standardized scale of Sign-Significate Relations (S-S) assessment.
4. The child is able to cooperate with the completion of TMS treatment and language assessment and has no serious behavioral problems.
5. The guardian of the child understands the content of this study and voluntarily signs the written informed consent.

Exclusion Criteria:

* 1. history of epilepsy or convulsive seizures. 2. having metal implants in the skull (e.g. aneurysm clips, metal stents, etc.) and electronic devices such as pacemakers and cochlear implants in the body.

  3. other serious neurological conditions that may affect language function (e.g., cerebral palsy, progressive neurological disorders, etc.).

  4. have a diagnosis of Autism Spectrum Disorder (ASD). 5. have a severe hearing or visual impairment. 6. participation in other clinical trials that may affect speech function. 7. breakage or infection at the scalp treatment site. 8.the fontanelle has not yet closed. 9. previous rTMS treatment in the last 3 months. 10. developmental quotient < 40 in any developmental domains; other circumstances that prevented cooperation with the study.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2026-01-16 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Language Developmental Quotient (DQ) via Gesell Developmental Schedules | Baseline (Day 0), Week 2 (End of intervention), and Week 4 (Follow-up).
  The language subscale of the Gesell Developmental Schedules is used to evaluate a child's language development. The result is expressed as a Developmental Quotient (DQ), a continuous score where 100 represents performance at the exact chronological age level. A higher DQ indicates better language abilities.

SECONDARY OUTCOMES:
Change from Baseline in Language Developmental Stage via Sign-Significate Relations (S-S) Assessment | Baseline (Day 0), Week 2 (End of intervention), and Week 4 (Follow-up).
  The S-S method is a standardized tool for the detailed diagnosis and classification of language developmental delay in children. It assesses both language comprehension and expression abilities, assigning the child to a specific developmental stage.The core outcome is the assigned Stage (I to V, with subdivisions). Higher stages indicate more advanced language development. For analysis, stages are often converted to an ordinal numerical score (e.g., Stage I=1, Stage II=2, etc.). The minimum score is 1 (lowest stage), and the maximum is 5 (highest stage).
Number of Participants with the Systematic Assessment for Treatment of Emergent Events (SAFTEE) [Safety and Tolerability] | From the start of intervention (Day 1) through the final follow-up (Week 4).
  Safety will be assessed by recording the incidence and severity of all adverse events (AEs) reported during the study. AEs include but are not limited to: headache, dizziness, scalp discomfort, tinnitus, irritability, and seizures. Severity will be graded as mild, moderate, or severe.

CONTACTS AND LOCATIONS:
Overall Officials: Fangkun Liu, MD, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangxi Autonomous Prefecture People's Hospital, The intersection of Century Avenue and Jianxin Road in Qianzhou Sub-district, Jishou (416000), Hunan, China., Jishou, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided